CLINICAL TRIAL: NCT02971345
Title: Endovascular Brachytherapy Combined With Stent Placement and Transcatheter Arterial Chemoembolization (TACE) for Treatment of HCC With Main Portal Vein Tumor Thrombus Versus TACE Alone: a Prospective Randomized Controlled Multicentre Trial
Brief Title: Endovascular Brachytherapy Combined With Stent Placement and TACE for HCC With Main Portal Vein Tumor Thrombus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Ruijin Hospital (Other); RenJi Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); The First Affiliated Hospital of Soochow University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Lishui Country People's Hospital (Other); Zhejiang University (Other); Changhai Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); The First Affiliated Hospital of Anhui Medical University (Other); The Second People's Hospital of Yibin (Other); The First Affiliated Hospital of Shanxi Medical University (Other); LanZhou University (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Hospital of China Medical University (Other); Fujian Medical University Union Hospital (Other); Fujian Provincial Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); ZhuHai Hospital (Other); Zhongshan Hospital Xiamen University (Other); Yancheng Third People's Hospital (Unknown); Changzhou Wujin People's Hospital (Unknown); Tengzhou Central People's Hospital (Other Government); Harbin Medical University (Other); Hunan Cancer Hospital (Other); First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZS-IR-2016
Record Dates: First submitted 2016-11-20; First posted 2016-11-22 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Tumor Thrombus
Keywords: Hepatocellular carcinoma; main portal vein tumor thrombus; endovascular brachytherapy; stent; chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Stents; Epirubicin; Ethiodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endovascular Brachytherapy&Stent&TACE (Experimental): Transarterial chemoembolization (TACE) is performed immediately following Iodine-125 seed strand and stent implantation.
  Epirubicin,ultra-fluid lipiodol and gelatin sponge articles are used in TACE.
  Interventions: Procedure: Stent and Iodine-125 seed strand implantation; Device: Stent; Device: Iodine-125 seed; Drug: Epirubicin; Drug: Ultra-fluid lipiodol; Other: Gelatin sponge articles
- TACE alone (Active Comparator): Only TACE is performed. Epirubicin, ultra-fluid lipiodol and gelatin sponge articles are used in TACE.
  Interventions: Drug: Epirubicin; Drug: Ultra-fluid lipiodol; Other: Gelatin sponge articles

INTERVENTIONS:
Procedure: Stent and Iodine-125 seed strand implantation — The patent second-order branch of the intrahepatic portal vein was punctured with a 22-gauge Chiba needle under ultrasound guidance.Stent and Iodine-125 seed strand are implanted by two 0.035-inch,150-cm-long wire.
  Arms: Endovascular Brachytherapy&Stent&TACE
Device: Stent — Bare stent should be placed through a 7-F, 23-cm-long sheath over the wire.
  Arms: Endovascular Brachytherapy&Stent&TACE
Device: Iodine-125 seed — The number of Iodine-125 seeds planned to be implanted was calculated by the following formula: N = length of obstructed main portal vein (mm)/4.5 + 4. These seeds were arranged linearly and sealed into a 4-F catheter continuously to construct a Iodine-125 seed strand.
  Arms: Endovascular Brachytherapy&Stent&TACE
Drug: Epirubicin — Epirubicin is a chemotherapy drug used in transarterial chemoembolization (TACE).Dosage: Epirubicin 30-60 mg per patient,depending on the situation of the patient.
Drug: Ultra-fluid lipiodol — Ultra-fluid lipiodol is a kind of embolization material used in TACE. Standard: 38% ultra-fluid lipiodol .
  Other Names: lipiodol
Other: Gelatin sponge articles — Gelatin sponge articles embolization material used in TACE. Standard: 350-560 um in diameter.

SUMMARY:
It is a prospective and multi-center clinical research in China to compare the efficacy, safety and related impact factors between TACE alone and endovascular brachytherapy combined with stent placement and TACE for HCC with main portal vein tumor thrombus.

DETAILED DESCRIPTION:
It is an open random prospective phase III clinical trial conducted by Principal Investigator Professor Zhi-ping Yan.Investigators in twenty-seven hospitals in China participate in.Patients with unresectable HCC with main portal vein tumor thrombus are enrolled. The investigators propose to recruitment 253 patients who are randomly assigned into the combined group (treated with endovascular brachytherapy combined with stent placement and TACE) and the control group (treated with TACE alone).There are 127 patients in combined group and 126 patients in control group. The criteria of inclusion and exclusion, and the methods of lab tests, imaging modality and treatment procedures are the same.

ELIGIBILITY:
Inclusion Criteria:

* (1) Hepatocellular carcinoma(HCC) diagnosis confirmed by needle biopsy or by two coincidental imaging techniques associated with increased α-fetoprotein according to the American Association for the Study of Liver Diseases (AASLD) guidelines;
* (2) According to the Barcelona Clinic Liver Cancer staging classification, HCC was unsuitable for resection, liver transplantation or percutaneous radiofrequency ablation;
* (3) Tumor thrombus, a low-attenuation intraluminal filling defect extending from intrahepatic portal vein branches adjacent to primary tumor into main portal vein, was confirmed by contrast-enhanced abdominal computer tomography (CT) or magnetic resonance imaging (MRI)
* (4) At least the first-order branch of the intrahepatic portal vein was patent in one lobe;
* (5) Child-Pugh classification grade A or B;
* (6) Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or less;

Exclusion Criteria:

* (1) Patients had a history of any therapy for HCC or portal vein tumor thrombus;
* (2) Advanced liver disease (bilirubin levels >3 mg/dL, Aspartate transaminase or Alanine aminotransferase >5 × upper limit of normal)；
* (3) Tumor invade the Inferior Vena Cava, extrahepatic spread;
* (4) Any contraindication to an arterial procedure such as impaired clotting tests (platelet count below 50 × 109/L or prothrombin activity below 50 %);
* (5) Renal failure,cardiac ejection fraction (<50 %) or end-stage disease;
* (6) Patients who were not capable of cooperation during the procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From the date of randomization until the date of death from any cause, assessed up to 24 months

SECONDARY OUTCOMES:
Time To Progression | From the date of first procedure of TACE or combined therapy until the time when the disease progresses from an intermediate to an advanced stage as defined by specific events, assessed up to 24 months
  Time to progression follow-up is done at three months interval after lesions defined as stable with treatment of TACE or combined therapy six months after enrollment until lesions are defined as disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiping Yan, MD, Principal Investigator — Department of Interventional Radiology, Zhongshan Hospital, Fudan University; Jianjun Luo, MD, Study Director — Department of Interventional Radiology, Zhongshan Hospital, Fudan University
Locations (1):
- Department of Interventional Radiology, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Luo J, Yan Z, Liu Q, Qu X, Wang J. Endovascular placement of iodine-125 seed strand and stent combined with chemoembolization for treatment of hepatocellular carcinoma with tumor thrombus in main portal vein. J Vasc Interv Radiol. 2011 Apr;22(4):479-89. doi: 10.1016/j.jvir.2010.11.029. PMID 21463757
- [Result] Luo JJ, Zhang ZH, Liu QX, Zhang W, Wang JH, Yan ZP. Endovascular brachytherapy combined with stent placement and TACE for treatment of HCC with main portal vein tumor thrombus. Hepatol Int. 2016 Jan;10(1):185-95. doi: 10.1007/s12072-015-9663-8. Epub 2015 Sep 4. PMID 26341514
- [Result] Yang M, Fang Z, Yan Z, Luo J, Liu L, Zhang W, Wu L, Ma J, Yang Q, Liu Q. Transarterial chemoembolisation (TACE) combined with endovascular implantation of an iodine-125 seed strand for the treatment of hepatocellular carcinoma with portal vein tumour thrombosis versus TACE alone: a two-arm, randomised clinical trial. J Cancer Res Clin Oncol. 2014 Feb;140(2):211-9. doi: 10.1007/s00432-013-1568-0. Epub 2013 Dec 28. PMID 24374800